CLINICAL TRIAL: NCT01325857
Title: Analgesic Efficacy of Bilateral Superficial Cervical Plexus Block in Robot-assisted Endoscopic Thyroidectomy Using a Transaxillary Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2010-0668
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group B (Experimental): Group B = Nerve block group
  Interventions: Procedure: Bilateral superficial cervical plexus block
- Group L (Placebo Comparator): Group L = Local wound infiltration group
  Interventions: Procedure: placebo
- Group C (Active Comparator): Group C = Control group
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Bilateral superficial cervical plexus block — Bilateral superficial cervical plexus block with 0.525% ropivacaine 20ml
  Arms: Group B
Procedure: placebo — Procedure: Bilateral superficial cervical plexus block with normal saline 20ml
  Arms: Group L
Procedure: Control group — Procedure: Local anesthetic infiltration at incision site with 0.525% ropivacaine 20ml
  Arms: Group C

SUMMARY:
This study was designed to investigate the analgesic effect of bilateral superficial cervical plexus block in patients undergoing robot-assisted endoscopic thyroidectomy. The investigators hypothesized that bilateral superficial cervical plexus blockade would reduce the patient's pain score by more than 10 (on a VAS scale of 0~100) compared to a placebo group and control group.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1 or 2 adult patients scheduled for robot-assisted endoscopic thyroidectomy

Exclusion Criteria:

* Patient refusal
* Bleeding diathesis
* Allergies to local anesthetics
* Patient unable to read consent form (Foreigner, illiterate)
* Pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score | Immediate post-operation (at recovery room) (day 1)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin S, Chung WY, Jeong JJ, Kang SW, Oh YJ. Analgesic efficacy of bilateral superficial cervical plexus block in robot-assisted endoscopic thyroidectomy using a transaxillary approach. World J Surg. 2012 Dec;36(12):2831-7. doi: 10.1007/s00268-012-1780-0. PMID 22956016